CLINICAL TRIAL: NCT03957824
Title: PRospEctiVE Study on implaNTable cardIOverter Defibrillator Therapy and SuddeN Cardiac Death in Adults With Congenital Heart Defects
Brief Title: PREVENTION-ACHD Risk Score
Acronym: PREVENTIONACHD
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Joris R. de Groot, Professor of Cardiac Electrophysiology and Atrial Fibrillation, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2014_248#C20141535
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Death, Sudden, Cardiac; Ventricular Fibrillation; Ventricular Tachycardia; Congenital Heart Disease
Keywords: Risk score; Risk prediction; Prevention
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia, Ventricular; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PREVENTION-ACHD risk score — The predicted risk of sudden cardiac death according to a risk score will be tested by the actual rate of sudden cardiac death

SUMMARY:
Sudden cardiac death (SCD) is one of the major causes of mortality in adults with congenital heart disease (ACHD). Risk stratification for sudden cardiac death in this patient group is challenging and at the current moment there are no clear guidelines on implantable cardioverter-defibrillator (ICD) implantation for primary prevention of SCD in this young patient population. The reason for this is the fact that this is a heterogenous group of patients and SCD is a relatively rare event. Because of this there have been no prospective studies on SCD in ACHD. However, multiple retrospective studies on ICD implantation in ACHD have shown that this treatment does appear to be effective. Researchers from the Academic Medical Center have identified several risk factors for sudden cardiac death. A risk score was created using this data, which has been validated in an internal and external cohort in a retrospective setting. The design of this study, including the conception of the risk score, its calculation method and validation will be published in an international scientific peer-reviewed journal.

The hypothesis of this study is that the risk score accurately predicts the risk of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* adult (≥18 years old) patient with a diagnosis of a congenital heart defect.

Exclusion Criteria:

* Patients of whom follow up is not possible, e.g. no permanent home address, living outside of or expecting to move out of the area wherein travelling to the investigating hospital outpatient clinic is possible.

  * Patients with documented sustained ventricular tachycardia or ventricular fibrillation.
  * Patients for whom the risk is not calculable because of a congenital heart disease diagnose not represented in the risk score.
  * Patients for whom the risk score is not calculable because of missing data
  * Patients with recent (<3 months ago) myocardial infarction.
  * Patients in whom the high SCD-risk status depends on an impaired ejection fraction that is expected to improve, e.g. due to tachycardiomyopathy.
  * Patients with a guideline defined contraindication for ICD implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with congenital heart disease with a diagnosis of one of the congenital heart defects displayed in the risk score model.
Sampling Method: Non-Probability Sample
Enrollment: 783 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Sudden cardiac death and ventricular fibrillation or sustained ventricular tachycardia | 2 years
  The rate of sudden cardiac death and ventricular fibrillation or sustained ventricular tachycardia in adult congenital heart disease patients

SECONDARY OUTCOMES:
Sudden cardiac death | 2 years
  The rate of sudden cardiac death in adult congenital heart disease patients

CONTACTS AND LOCATIONS:
Overall Officials: Joris R de Groot, MD, PhD, Principal Investigator — Academic Medical Center - University of Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vehmeijer JT, Koyak Z, Zwinderman AH, Harris L, Peinado R, Oechslin EN, Silversides CK, Bouma BJ, Budts W, van Gelder IC, Oliver JM, Mulder BJM, de Groot JR. PREVENTION-ACHD: PRospEctiVE study on implaNTable cardioverter-defibrillator therapy and suddeN cardiac death in Adults with Congenital Heart Disease; Rationale and Design. Neth Heart J. 2019 Oct;27(10):474-479. doi: 10.1007/s12471-019-1297-3. PMID 31270738